CLINICAL TRIAL: NCT01349322
Title: A Phase III Trial of Accelerated Whole Breast Irradiation With Hypofractionation Plus Concurrent Boost Versus Standard Whole Breast Irradiation Plus Sequential Boost for Early-Stage Breast Cancer
Brief Title: Higher Per Daily Treatment-Dose Radiation Therapy or Standard Per Daily Treatment Radiation Therapy in Treating Patients With Early-Stage Breast Cancer That Was Removed by Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-1005; NCI-2011-02669 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000700069; NCT03553797 (obsolete NCT alias)
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Results first posted 2023-04-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole breast irradiation + sequential boost (Active Comparator): Standard fractionation whole breast irradiation (WBI) with sequential boost.
  Interventions: Radiation: Standard fractionation whole breast irradiation; Radiation: Sequential boost
- Hypofractionated whole breast irradiation + concurrent boost (Experimental): Hypofractionated whole breast (H-WBI) irradiation with a concurrent boost
  Interventions: Radiation: Hypofractionated whole breast irradiation; Radiation: Concurrent boost

INTERVENTIONS:
Radiation: Standard fractionation whole breast irradiation — Target-based radiation using three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) to deliver 25 fractions of 2.0 Gy for a total dose of 50.0 Gy or 16 fractions of 2.67 Gy for a total dose of 42.7 Gy. Must begin within 9 weeks of last surgery or chemotherapy delivery.
  Other Names: three-dimensional conformal radiation therapy (3D-CRT); intensity-modulated radiation therapy (IMRT)
  Arms: Whole breast irradiation + sequential boost
Radiation: Hypofractionated whole breast irradiation — Target-based radiation using three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) to deliver 15 fractions of 2.67 Gy for a total dose of 40.0 Gy. Must begin within 9 weeks of last surgery or chemotherapy delivery.
  Other Names: three-dimensional conformal radiation therapy (3D-CRT); intensity-modulated radiation therapy (IMRT)
  Arms: Hypofractionated whole breast irradiation + concurrent boost
Radiation: Concurrent boost — 15 fractions of 3.2 Gy for a total dose of 48 Gy to the lumpectomy cavity. Given concurrently with treatment to the entire breast. May be given by either electron beam or photon beams using either 3D-CRT or IMRT.
  Arms: Hypofractionated whole breast irradiation + concurrent boost
Radiation: Sequential boost — 6 fractions of 2.0 Gy per fraction for a total dose of 12 Gy or 7 fractions of 2.0 Gy for a total dose of 14 Gy to the lumpectomy cavity. May be given by either electron beam or photon beams using either 3D-CRT or IMRT. Begins without a treatment break after completion of the treatment to the entire breast.
  Arms: Whole breast irradiation + sequential boost

SUMMARY:
RATIONALE: It is not yet know whether higher per daily radiation therapy is equally as effective as standard per daily radiation therapy in treating breast cancer.

PURPOSE: This randomized phase III trial studies how well an accelerated course of higher per daily radiation therapy with concomitant boost works compared to standard per daily radiation therapy with a sequential boost in treating patients with early-stage breast cancer that was removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether an accelerated course of hypofractionated whole-breast irradiation (WBI) including a concomitant boost to the tumor bed in 15 fractions following lumpectomy will prove to be non-inferior in local control to a regimen of standard WBI with a sequential boost following lumpectomy for early-stage breast cancer patients.

Secondary

* To determine whether breast-related symptoms and cosmesis from accelerated WBI that is hypofractionated (in only 3 weeks) with a concomitant boost is non-inferior to standard WBI with sequential boost.
* To determine whether the risk of late cardiac toxicity in patients with left-sided breast cancer treated with hypofractionation will be non-inferior to conventional fractionated radiation therapy (RT) based upon analysis of radiation dosimetry from CT-based treatment planning and normal tissue complication probability (NTCP) calculations.
* To determine whether CT-based conformal methods intensity-modulated radiation therapy (IMRT) and three-dimensional conformal radiotherapy (3D-CRT) for WBI are feasible in a multi-institutional setting following lumpectomy in early-stage breast cancer patients and whether dose-volume analyses can be established to assess treatment adequacy and likelihood of toxicity.
* To determine that cosmetic results and breast-related symptoms 3 years after hypofractionated breast radiation with concomitant boost will not be inferior to that obtained 3 years after WBI with sequential boost.
* To determine whether future correlative studies can identify individual gene expressions and biological host factors associated with toxicity and/or local recurrence from standard and hypofractionated WBI.
* If shown to be non-inferior, to then determine if accelerated course of hypofractionated WBI including a concomitant boost to the tumor bed in 15 fractions following lumpectomy will prove to be superior in local control to a regimen of standard WBI with a sequential boost following lumpectomy for early-stage breast cancer patients.
* To determine whether treatment costs for hypofractionated WBI with concomitant boost are not higher than WBI with sequential boost.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 50 vs. ≥ 50 years), prior chemotherapy (yes vs. no), estrogen-receptor status (+ vs. -), and histology grade (1-2 vs. 3). Patients are randomized to 1 of 2 treatment arms. Treatment begins within 9 weeks of last surgery or chemotherapy delivery.

After completion of study therapy, patients are followed at 1 month, at 6 months, and then yearly.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically proven diagnosis of breast cancer resected by lumpectomy and whole breast irradiation with boost without regional nodal irradiation planned
2. The patient must be female
3. The patient must meet at least one of the three following criteria:

   * A. Pathological stage I, II Breast Cancer AND at least one of the following:

     * Age < 50 years or
     * Positive axillary nodes or
     * Lymphovascular space invasion or
     * 2 or more close resection margins (> 0 mm to ≤ 2 mm) or
     * 1 close resection margin and extensive intraductal component (EIC) [Per College of American Pathologist (CAP) Recommendation] or
     * Focally positive resection margins or
     * Non-hormone sensitive breast cancer (estrogen receptor (ER)- and progesterone receptor(PR)-negative) or
     * Grade III histology or
     * Oncotype recurrence score > 25 or
   * B. Pathological stage 0 breast cancer with nuclear grade 3 ductal carcinoma in situ (DCIS) and patient age <50 years or
   * C. Post-neoadjuvant pathological 0, I, II breast cancer resected by lumpectomy after neoadjuvant systemic therapy
4. Study entry must be within 50 days from whichever comes later: last surgery (breast or axilla) or last chemotherapy. The day of surgery is Day "0".
5. If multifocal breast cancer, then it must have been resected through a single lumpectomy incision with negative margins
6. Breast-conserving surgery with margins defined as follows: (also see 3.1.3 for eligibility)

   * Negative margins defined as no tumor at the resected specimen edge.
   * Close resection margins > 0 mm to ≤ 2 mm. as follows:

     * One close resection margin and EIC (per College of American Pathologist (CAP) Recommendation)
     * 2 or more close resection margins.
   * A focally positive resection margin
7. For invasive breast cancer the axilla must be staged by one of the following:

   * Sentinel node biopsy alone, if sentinel node is negative, i.e. any of the following:

     * pN0: no regional lymph node metastasis identified histologically,
     * pN0(i-): pN0 and immunohistochemical (IHC) negative, or
     * pN0(i+): pN0 and IHc positive;
   * Sentinel node biopsy alone, OR followed by axillary node dissection per investigator discretion, for clinically node negative patients as described below:

     * microscopic sentinel node positive (pN1mic)
     * one or two sentinel nodes positive (pN1) without extracapsular extension
     * negative sentinel node biopsy after neoadjuvant chemotherapy
   * Axillary node dissection is required following sentinel node (SN) biopsy with a minimum total of 6 axillary nodes if any of the following exist:

     * for > 2 positive SN
     * any positive SN biopsy after neoadjuvant chemotherapy
     * for clinically (by either imaging or examination) T3 disease
     * for extracapsular extension
   * Axillary dissection alone (with a minimum of 6 axillary nodes)
8. Age ≥ 18
9. CT-imaging of the ipsilateral breast within 28 days prior to study entry for the radiation treatment planning. Must be able to delineate on CT scan the extent of the target lumpectomy cavity for boost
10. Appropriate stage for protocol entry, including no clinical evidence for distant metastases, based upon the following minimum diagnostic workup:

    * History/physical examination, including breast exam (inspection and palpation of the breasts) and documentation of weight and Zubrod Performance Status of 0-2 within 28 days prior to study entry;
    * Right and left mammography within 90 days of diagnostic biopsy establishing diagnosis
11. Patients must have had ER analysis performed on the primary breast tumor prior to study entry according to current American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) Guideline Recommendations for hormone receptor testing. If negative for ER, assessment of PR must also be performed according to current ASCO/CAP Guideline Recommendations for hormone receptor testing (http://www.asco.org)
12. Complete blood count (CBC)/differential obtained within 14 days prior to study entry, with adequate bone marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
    * Platelets ≥ 75,000 cells/mm3
    * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
13. Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days of study entry
14. Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during radiation therapy
15. Patient must provide study specific informed consent prior to study entry
16. Breast implants allowed

Exclusion criteria:

1. American Joint Committee on Cancer (AJCC) pathologic T4, N2 or N3, M1 pathologic stages III or IV breast cancer
2. Treatment plan that includes regional node irradiation
3. Prior invasive non-breast malignancy (except non-melanomatous skin cancer, carcinoma in situ of the cervix) unless disease free for a minimum of 5 years prior to study entry
4. Prior invasive or in-situ carcinoma of the breast [-prior lobular carcinoma in situ (LCIS) is eligible]
5. Two or more breast cancers not resectable through a single lumpectomy incision
6. Bilateral breast cancer
7. DCIS only (without an invasive component) and age ≥ 50 years
8. DCIS nuclear grade 1 or 2 only (without an invasive component) and age < 50 years
9. Invasive breast cancer and low risk for 5-year in breast recurrence after lumpectomy with negative margins that does not meet one of the eligibility factors in 3.1.3.
10. Unable to delineate on CT scan the extent of the target lumpectomy cavity for boost (Placement of surgical clips to assist in treatment planning of the boost is strongly recommended, see Section 6.4.2 for details)
11. Suspicious unresected microcalcification, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign
12. Non-epithelial breast malignancies such as sarcoma or lymphoma
13. Paget's disease of the nipple
14. Male breast cancer
15. Prior radiotherapy to the breast or prior radiation to the region of the ipsilateral breast that would result in overlap of radiation therapy fields
16. Intention to administer concurrent chemotherapy for current breast cancer.
17. Severe, active co-morbidity, defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    * Transmural myocardial infarction within the last 6 months
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration;
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive
18. Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
19. Active systemic lupus, erythematosus, or any history of scleroderma, dermatomyositis with active rash
20. Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2354 (Actual)
Dates: Start 2011-05-24 (Actual); Primary Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Vicini, MD, FACR, Principal Investigator — St. Joseph Mercy Oakland; Gary M. Freedman, MD, Study Chair — University of Pennsylvania; Julia R. White, MD, Study Chair — Ohio State University; Douglas W. Arthur, MD, Study Chair — Virginia Commonwealth University
Locations (415):
- United States (386):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - 21st Century Oncology-Scottsdale, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - 21st Century Oncology - El Segundo, El Segundo, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - 21st Century Oncology - Fort Walton Beach, Fort Walton Beach, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Cancer Center of Putnam, Palatka, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The Villages Regional Hospital, The Villages, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - IU Health West Hospital, Avon, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - GenesisCare USA - Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - GenesisCare USA - Farmington Hills, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - KCC Radiation Oncology at Monroe Cancer Center, Monroe, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Ocean Medical Center, Brick, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Saint Peter's Health Partners, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Cayuga Medical Center, Ithaca, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - The Coleman Radiation Center-Carteret General Hospital, Morehead City, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - NHRMC Radiation Oncology - 16th Street, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Rockingham Memorial Hospital Hahn Cancer Center, Harrisonburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Harrison Medical Center, Bremerton, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Beloit Memorial Hospital, Beloit, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (20):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - Irving Greenberg Family Cancer Centre, Ottawa, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Litwinsky
- Shizuoka Cancer Center, Shizuoka, Suntou, Japan
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (2):
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Yonsei University Health System-Severance Hospital, Seoul
- Kantonsspital Aarau, Aarau, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Started | 1169 | 1185
Eligible Population | 1124 | 1138
Adverse Event Population (Eligible participants who started protocol treatment and had adverse event data) | 1100 | 1123
Quality of Life Population (Eligible, consented, and accrued when QOL substudy was open to enrollment) | 429 | 449
Completed | 1124 | 1138
Not Completed | 45 | 47
Not completed — Protocol Violation | 45 | 47

BASELINE CHARACTERISTICS:
Population: Eligible population
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost | Total
Number analyzed (Participants) | 1124 | 1138 | 2262
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [47 to 64] | 55 [47 to 64] | 55 [47 to 64]
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 403 | 400 | 803
  ≥ 50 years | 721 | 738 | 1459
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1124 | 1138 | 2262
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 72 | 129
  Not Hispanic or Latino | 1046 | 1051 | 2097
  Unknown or Not Reported | 21 | 15 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 16
  Asian | 65 | 62 | 127
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 135 | 131 | 266
  White | 887 | 909 | 1796
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 24 | 19 | 43
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 896 | 943 | 1839
    1 | 222 | 190 | 412
    2 | 6 | 5 | 11
Resection Margin Status [Count of Participants; unit: Participants]
  Negative margins (no tumor at the resected specimen edge) | 942 | 942 | 1884
  Close resection margins (>0mm to ≤2mm / Focally positive resection margin) | 182 | 196 | 378
Axillary Staging Method [Count of Participants; unit: Participants]
  Sentinel node biopsy alone | 883 | 934 | 1817
  Sentinel node biopsy alone or followed by axillary node dissection | 183 | 163 | 346
  Sentinel node biopsy followed by axillary dissection/minimum 6 axillary nodes | 13 | 11 | 24
  Axillary dissection alone (with a minimum 6 axillary nodes) | 30 | 22 | 52
  None: non-invasive breast cancer | 15 | 8 | 23
Radiation Therapy Technique (plan at randomization) [Count of Participants; unit: Participants]
  3D-CRT | 887 | 888 | 1775
  IMRT | 237 | 250 | 487
Received Chemotherapy [Count of Participants; unit: Participants]
  Yes | 678 | 697 | 1375
  No | 446 | 441 | 887
Estrogen receptor (ER) Status [Count of Participants; unit: Participants]
  Negative | 335 | 350 | 685
  Positive | 789 | 788 | 1577
Histologic Grade [Count of Participants; unit: Participants] — A histologic measure of how closely a cancer cell nucleus resembles that of a normal cell, or a measure of how abnormal a cancer nuclear is. It is generally graded as 1 (resembles normal), 2 (moderately abnormal), and 3 (markedly abnormal).
  Participants
    1-2 | 535 | 545 | 1080
    3 | 589 | 593 | 1182
Pathologic Stage [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 7th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. The higher the number after the N, the greater the involvement of regional lymph nodes. M0 indicates no distant metastasis.
  Participants
    Stage 0 (Tis, N0, M0) | 36 | 34 | 70
    Stage I (T1/T1mi, N0, M0 or T0/T1/T1mi, N1mi, M0) | 683 | 727 | 1410
    Stage II (T0/T1/T1mi, N1, M0 or T2, N0, M0 or T2, N1, M0 or T3, N0, M0) | 399 | 376 | 775
    Stage III (T0/T1/T1mi/T2, N2, M0 or T3, N1/N2, M0 or T4, N0/N1/N2, M0 or Any T,N3,M0) | 2 | 0 | 2
    Stage IV (Any T, Any N, M1) | 4 | 1 | 5
Oncotype recurrence score > 25 [Count of Participants; unit: Participants] — An oncotype recurrence score comes from an analysis of a sample of a cancer tumor to see the activity of certain genes that can affect the cancer's outcome and how likely it is to grow and spread. A score >25 means you have a higher risk that the disease might come back. Both hormone treatment and chemotherapy are likely to be recommended.
  Participants
    No | 1030 | 1014 | 2044
    Yes | 94 | 124 | 218
Pathologic stage 0 breast cancer wtih nuclear grade 3 DCIS and patient age <50 years [Count of Participants; unit: Participants] — DCIS: Ductal carcinoma in situ
  Participants
    No | 1092 | 1107 | 2199
    Yes | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With In-breast Recurrence (Local Failure)
Description: In-breast recurrence (IBR) is defined as any of the following: invasive local recurrence-ipsilateral breast (within treatment field); invasive local recurrence-ipsilateral breast (outside treatment field); non-invasive local recurrence-ipsilateral breast (within treatment field); or non-invasive local recurrence-ipsilateral breast (outside treatment field). Time to IBR is defined as time from randomization to the date of first IBR, last known follow-up (censored), or death without IBR (competing risk). IBR rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. 5-year rates are provided.
Time Frame: From randomization to last follow-up. Evaluated weekly during radiation therapy (RT), last day of RT, 1, 6, and 12 months after RT completion, then annually. Maximum follow-up at time of analysis was 10.1 years. Five-year rates are reported here.
Population: Eligible population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Whole Breast Irradiation + Sequential Boost (Arm 1): Standard fractionation whole breast irradiation (WBI) with sequential boost.
  Standard fractionation whole breast irradiation: Target-based radiation using three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) to deliver 25 fractions of 2.0 Gy for a total dose of 50.0 Gy or 16 fractions of 2.67 Gy for a total dose of 42.7 Gy. Must begin within 9 weeks of last surgery or chemotherapy delivery.
  Sequential boost: 6 fractions of 2.0 Gy per fraction for a total dose of 12 Gy or 7 fractions of 2.0 Gy for a total dose of 14 Gy to the lumpectomy cavity. May be given by either electron beam or photon beams using either 3D-CRT or IMRT. Begins without a treatment break after completion of the treatment to the entire breast.
- Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2): Hypofractionated whole breast (H-WBI) irradiation with a concurrent boost
  Hypofractionated whole breast irradiation: Target-based radiation using three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) to deliver 15 fractions of 2.67 Gy for a total dose of 40.0 Gy. Must begin within 9 weeks of last surgery or chemotherapy delivery.
  Concurrent boost: 15 fractions of 3.2 Gy for a total dose of 48 Gy to the lumpectomy cavity. Given concurrently with treatment to the entire breast. May be given by either electron beam or photon beams using either 3D-CRT or IMRT.
Arm/Group | Whole Breast Irradiation + Sequential Boost (Arm 1) | Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2)
Number analyzed (Participants) | 1124 | 1138
percentage of participants | 2.0 [1.4 to 2.9] | 1.9 [1.3 to 2.7]
Statistical Analysis 1: Comparison: Whole Breast Irradiation + Sequential Boost (Arm 1) vs Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2); Assuming Arm 1 5-year IBR of 1.59%, for hypothesized upper bound hazard ratio (HR) of 2.12 (Arm 2 5-year IBR of 3.33%), 46 IBR events provide >80% power to conclude non-inferiority with one-sided significance level = 0.05. Null hypothesis: HR ≥ 2.12 (inferior). Alternative hypothesis: HR < 2.12 (non-inferior). See "Limitations and Caveats" section; Test type: Non-Inferiority — Non-inferiority is defined as a hazard ratio upper limit of 2.12; p = 0.039, Regression, Cox; Hazard Ratio (HR) = 1.32, 90% CI 2-sided [0.84 to 2.05] — Cause-specific hazard ratio; reference level = Arm 1

2. Secondary Outcome: Percentage of Participants Alive
Description: Failure is defined as death due to any cause. Failure time (overall survival time) is defined as the time from randomization to the date of death or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method and distributions between the two arms are compared using the log-rank test. Five-year rates are provided here.
Time Frame: From randomization to last follow-up. Evaluated weekly during radiation therapy (RT), last day of RT, 1, 6, and 12 months after RT completion, then annually. Maximum follow-up at time of analysis was 10.1 years. Five-year rates are provided here.
Population: Eligible population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Number analyzed (Participants) | 1124 | 1138
percentage of participants | 95.7 [94.4 to 96.9] | 95.1 [93.8 to 96.4]
Statistical Analysis 1: Comparison: Whole Breast Irradiation + Sequential Boost vs Hypofractionated Whole Breast Irradiation + Concurrent Boost; Test type: Superiority; p = 0.96, Log Rank — Two-sided significance level = 0.05

3. Secondary Outcome: Percentage of Participants Alive Without Disease
Description: Disease-free survival (DFS) time is defined as time from randomization to local-regional disease recurrence, distant metastases, second/new primary, death due to any cause or last known follow-up (censored). DFS rates are estimated by the Kaplan-Meier method and distributions between the two arms are compared using the log-rank test. Five-year rates are provided here.
Time Frame: as for outcome 2
Population: Eligible population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Number analyzed (Participants) | 1124 | 1138
percentage of participants | 90.2 [88.5 to 92.0] | 88.5 [86.7 to 90.4]
Statistical Analysis 1: Comparison: Whole Breast Irradiation + Sequential Boost vs Hypofractionated Whole Breast Irradiation + Concurrent Boost; Test type: Superiority; p = 0.14, Log Rank — Two-sided significance level = 0.05

4. Secondary Outcome: Percentage of Participants Alive Without Distant Disease
Description: Distant disease-free survival (DDFS) time is defined as time from randomization to distant metastases, second/new primary, death due to any cause or last known follow-up (censored). DDFS rates are estimated by the Kaplan-Meier method and distributions between the two arms are compared using the log-rank test. Five-year rates are provided here.
Time Frame: as for outcome 2
Population: Eligible population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Number analyzed (Participants) | 1124 | 1138
percentage of participants | 91.5 [89.9 to 93.2] | 90.2 [88.4 to 91.9]
Statistical Analysis 1: Comparison: Whole Breast Irradiation + Sequential Boost vs Hypofractionated Whole Breast Irradiation + Concurrent Boost; Test type: Superiority; p = 0.34, Log Rank — Two-sided significance level = 0.05

5. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported as Definitely, Probably, or Possibly Related to Protocol Treatment
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data
Time Frame: From randomization to last follow-up. Evaluated weekly during radiation therapy (RT), last day of RT, 1, 6, and 12 months after RT completion, then annually. Maximum follow-up at time of analysis was 10.1 years.
Population: Adverse event population
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Number analyzed (Participants) | 1100 | 1123
Participants
  Grade 1 | 427 | 554
  Grade 2 | 379 | 290
  Grade 3 | 34 | 35
  Grade 4 | 2 | 4
  Grade 5 | 0 | 0

6. Secondary Outcome: Change in Breast Cancer Treatment Outcome Scale (BCTOS) Cosmesis Subscale Score From Baseline to 3 Years
Description: The BCTOS cosmesis subscale score measures perceived aesthetic (e.g., breast shape) status . Patients rated each item using a four-point scale evaluating the differences between the treated and the untreated breast (1=no difference, 2=slight difference, 3=moderate difference, 4=large difference) with higher scores indicating a worse outcome. The score for each subscale is the mean of the ratings over all items belonging to that specific subscale. Change was calculated as the value at 3 years minus the value at baseline. A positive change reflects a decline at 3 years and a negative change reflects an improvement at 3 years.
Time Frame: Baseline and 3 years
Population: Quality of life population, with data at baseline and 3 years.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Whole Breast Irradiation + Sequential Boost (Arm 1) | Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2)
Number analyzed (Participants) | 254 | 274
score on a scale | 0.16 [0.08 to 0.24] | 0.18 [0.11 to 0.25]
Statistical Analysis 1: Comparison: Whole Breast Irradiation + Sequential Boost (Arm 1) vs Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2); Test type: Non-Inferiority — Null hypothesis (H0) of inferiority: the mean change in cosmetic subscale score in Arm 2 will be at least 0.4 standard deviations worse than in Arm 1. If H0 is rejected, then non-inferiority can be concluded; p < 0.0001, t-test, 1 sided — One-side significance level = 0.025; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.08 to 0.13], Standard Deviation 0.62

7. Secondary Outcome: Percentage of Participants With a Physician-reported Cosmetic Score of Excellent or Good at 3 Years
Description: Physicians rated cosmesis using a four point scale:
  * Excellent: When compared to the untreated breast or the original appearance of the breast, there is minimal/no difference in the size or shape of the treated breast.
  * Good: There is a slight difference in the size or shape of the treated breast as compared to the opposite breast or the original appearance of the treated breast.
  * Fair: Obvious differences in the size and shape of the treated breast. This change involves quarter or less of the breast.
  * Poor: Marked change in the appearance of the treated breast involving more than a quarter of the breast tissue.
Time Frame: 3 years
Population: Quality of life population, with data at 3 years.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Whole Breast Irradiation + Sequential Boost (Arm 1) | Hypofractionated Whole Breast Irradiation + Concurrent Boost (Arm 2)
Number analyzed (Participants) | 199 | 216
percentage of participants | 86 [80 to 90] | 82 [77 to 87]

8. Secondary Outcome: Correlation Between Dose-volume Data and Both Adverse Events and Efficacy
Time Frame: From randomization to end of follow-up.
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Translational Research of Single Nucleotide Polymorphisms (SNPs) in Transforming Growth Factor Beta 1 (TGFB1) and Ataxia-Telangiesctasia Mutated (ATM) Genes
Time Frame: From randomization to last follow-up.
Population: The protocol did not provide sufficient detail to meet current National Cancer Institute requirements for release of specimens from the NRG Oncology tissue bank for the protocol-specified analysis, therefore no assays were performed, and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Treatment Cost
Time Frame: From randomization to end of treatment.
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Weekly during radiation therapy (RT), last day of RT, 1, 6, and 12 months after RT completion, then annually. Maximum follow-up at time of analysis was 10.1 years.
Description: All-cause mortality was assessed in the eligible population. Adverse events were assessed in the adverse event population.
Arm/Group | Whole Breast Irradiation + Sequential Boost | Hypofractionated Whole Breast Irradiation + Concurrent Boost
All-Cause Mortality (participants affected / at risk) | 87/1124 | 86/1138
Serious Adverse Events (participants affected / at risk) | 18/1100 | 20/1123
Other Adverse Events (participants affected / at risk) | 866/1100 | 910/1123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Whole Breast Irradiation + Sequential Boost (N=1100) | Hypofractionated Whole Breast Irradiation + Concurrent Boost (N=1123)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Flu like symptoms (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Localized edema (General disorders) | 2 | 1
Pain (General disorders) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Hematoma (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Lymphedema (Vascular disorders) | 1 | 2
Peripheral ischemia (Vascular disorders) | 1 | 0
Visceral arterial ischemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Whole Breast Irradiation + Sequential Boost (N=1100) | Hypofractionated Whole Breast Irradiation + Concurrent Boost (N=1123)
Nausea (Gastrointestinal disorders) | 60 | 56
Fatigue (General disorders) | 435 | 427
Localized edema (General disorders) | 123 | 116
Pain (General disorders) | 160 | 144
Dermatitis radiation (Injury, poisoning and procedural complications) | 399 | 384
Arthralgia (Musculoskeletal and connective tissue disorders) | 116 | 124
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 58 | 69
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 67 | 82
Pain in extremity (Musculoskeletal and connective tissue disorders) | 69 | 62
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 123 | 105
Headache (Nervous system disorders) | 44 | 58
Peripheral sensory neuropathy (Nervous system disorders) | 72 | 85
Depression (Psychiatric disorders) | 43 | 57
Insomnia (Psychiatric disorders) | 58 | 77
Breast atrophy (Reproductive system and breast disorders) | 63 | 64
Breast pain (Reproductive system and breast disorders) | 325 | 320
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 89 | 109
Dry skin (Skin and subcutaneous tissue disorders) | 49 | 70
Erythema multiforme (Skin and subcutaneous tissue disorders) | 83 | 79
Pruritus (Skin and subcutaneous tissue disorders) | 125 | 86
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 191 | 172
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 464 | 458
Skin induration (Skin and subcutaneous tissue disorders) | 92 | 97
Hot flashes (Vascular disorders) | 204 | 190
Hypertension (Vascular disorders) | 84 | 67
Lymphedema (Vascular disorders) | 79 | 84

LIMITATIONS AND CAVEATS:
Due to a lower than anticipated incidence of in-breast recurrence (IBR), the protocol was amended to allow for timely reporting of the trial results with at least 46 IBR events, while maintaining statistical integrity and reflecting current knowledge of the observed IBR incidence in the control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01349322/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01349322/ICF_001.pdf